CLINICAL TRIAL: NCT05822427
Title: Long-term Follow-up of Study Participants Who Received an Allogeneic Chimeric Antigen Receptor T-Cell Product in an Imugene Ltd. Clinical Study
Status: Recruiting | Type: Observational
Sponsor: Imugene Limited (Industry)
Responsible Party: Sponsor
Other Study IDs: PBCAR-LTF
Record Dates: First submitted 2023-04-10; First posted 2023-04-20 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Participants Who Received an Allogeneic Chimeric Antigen Receptor T-Cell Product (PBCAR) in a Precision BioSciences, Inc., Clinical Study
Keywords: Allogeneic chimeric antigen receptor (CAR) T cell products; azer-cel

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Unless participants entering the study have three consecutive negative azer-cel persistence tests results when entering the study, participants will undergo persistence testing whilst on study untill three consecutive negative tests are confirmed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The goal of this observational study is to collect information on the long-term safety of study participants who received an Allogeneic Chimeric Antigen Receptor (CAR) T-Cell Product in an Imugene Clinical Study. The main questions it aims to answer are:

* What are the frequency, severity, duration, and outcome of clinically significant Clinical Events of Interest (CEI)?
* What is the duration of response and overall survival time after taking an allogeneic CAR T-Cell product on an Imugene clinical study?

Participants will have a yearly visit either face to face or remotely for up to 15 years to check for CEI.

DETAILED DESCRIPTION:
This is a Long-Term Follow-Up (LTFU) observational study designed primarily to collect data regarding CEI for up to 15 years following participation in an Imugene clinical study for subjects who received azer-cel. This study protocol does not include administration of azer-cel; however, subjects may receive standard of care treatment or investigational products other than azer-cel through participation in other clinical studies during the period of this observational study.

ELIGIBILITY:
Inclusion Criteria:

* Receipt of at least 1 dose of azer-cel in an Imugene clinical study.
* A signed informed consent form (ICF).
* Willingness and ability to adhere to the study schedule and all other protocol requirements.

Exclusion Criteria:

* No unique exclusion criteria apply to this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any participant who has received a azer-cel in an Imugene clinical study can be enrolled into this LTFU study.
Sampling Method: Non-Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2020-08-25 (Actual); Primary Completion 2039-12 (Estimated); Study Completion 2039-12 (Estimated)

PRIMARY OUTCOMES:
Frequency of Clinically Significant Clinical Events of Interest (CEI) | Up to 15 years
Severity of Clinically Significant CEI | Up to 15 years
Duration of Clinically Significant CEI | Up to 15 years
Outcome of Clinically Significant CEI | Up to 15 years

SECONDARY OUTCOMES:
Duration of Disease Response | Up to 15 years
Overall Survival Rate | Up to 15 years
Azer-cel Persistence | Up to 15 years

CONTACTS AND LOCATIONS:
Locations (1):
- Science 37, Inc., Culver City, California, United States

IPD SHARING:
Plan to Share IPD: Undecided